CLINICAL TRIAL: NCT04886362
Title: Safety and Efficacy and of Ivermectin for the Prevention of Severe Disease in Patients With COVID-19: A Randomized, Controlled, Double-Blind Clinical Study.
Brief Title: Ivermectina Colombia (IVERCOL)
Acronym: IVERCOL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ayudas Diagnosticas Sura S.A.S (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVERCOL01
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pneumonia
Keywords: Ivermectin; COVID-19; Ambulatory
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Ivermectin 600 mcg/kg every 12 hours for 5 days.
  Interventions: Drug: Ivermectin
- Control Group (Placebo Comparator): Same volume like ivermectin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — Treatment with Ivermectin in the first 7 days from symptoms onset.
  Arms: Intervention Group
Drug: Placebo — Treatment with Placebo in the first 7 days from symptoms onset.
  Arms: Control Group

SUMMARY:
A parallel, prospective, double-blind, placebo-controlled clinical trial will be conducted in the population affiliated to EPS SURAMERICANA S.A. with positive test for antigen and PCR for SARS-CoV-2. Participants will be randomly assigned in a 1: 1 ratio to the intervention group or the control group using a sequence of random numbers. The patients included will be those with less than 7 days from the onset of symptoms, and without evidence of serious disease.

One group will be assigned oral ivermectin therapy at a dose of 600 mcg/kg every 12 hours for 5 consecutive days, and the other group will received placebo. A minimum sample size of 483 patients for each arm was calculated to observe differences. All randomized patients will be included in the analysis according to the randomization arm (intention-to-treat analysis).

The primary objective is to evaluate the efficacy of ivermectin in the prevention of severe disease, reduction in the rate of hospitalization, reduction of ICU stay, and mortality. This evaluation will be carried out up to 28 days after the intervention begins. Given the public health emergency, the study is expected to be completed in a period of 6 months from the INVIMA approval.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years.
* Patients with positive antigen test or RT-PCR for SARS-CoV-2.
* Patients with less than 7 days from symptoms onset.
* Patients with indication for outpatient management.
* Patients with mild disease according to the official guide "Pneumonia Diagnosis and Treatment Scheme for Novel Coronavirus Infection (Trial Version 8)": Subjects with mild symptoms, with or without radiological signs of pneumonia, with oxygen saturation>90% . - Able to provided consent to participate.

Exclusion Criteria:

* Patients who at the time of admission require hospitalization and / or supplemental oxygen.
* Known history of allergy to ivermectin.
* Known medical history of liver disease.
* Belong to another clinical trial evaluating the efficacy of an investigational drug against COVID-19.
* The following comorbidities:

  * Immunosuppression or HIV.
  * Acute or chronic kidney failure.
  * Current neoplasia.
* Currently use of warfarin, erdafitinib, or quinidine.
* Have received vaccination for SARS-CoV-2.
* Ivermectin consumption prior to inclusion in the research protocol.
* The patient does not accept the conditions of home care and monitoring.
* The patient desists from participating in the study.
* Women in pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 966 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Composite Outcome | 28 days
  Proportion of patients progressing to severe COVID-19. Progression to severe disease will be considered when at least one of the following clinical situations occurs (composite outcome) the first thing that occurs in each patient during the 28 days after the intervention begins:
  1. Hypoxemia (oxygen saturation ≤90%) and need for supplemental oxygen in home care program; or
  2. Need for hospitalization includes general bed, ICU or ICU; or
  3. Death from any cause.

SECONDARY OUTCOMES:
Hypoxemia (oxygen saturation ≤90%) and need for supplemental oxygen in home care program. | 28 days
Need for hospitalization including general bed, ICU or ICU. | 28 days
Death from any cause. | 28 days
Proportion of patients with 4 or more points on the WHO scale (8-point ordinal scale). | 28 days
Number of days with supplemental oxygen requirement. | 28 days
Number of days on ICU management. | 28 days
Number of days on endotracheal intubation (IOT). | 28 days
Number of days of hospitalization. | 28 days
Number and type of serious and non-serious adverse events. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Chacón Jimenez, MD, Study Director — Emergencies Department Director

IPD SHARING:
Plan to Share IPD: No
Data will be available on request and the proper approval from ethics committee.